CLINICAL TRIAL: NCT05718505
Title: Comparison of the Atmo Motility Gas Capsule System to the Reference Standard (SmartPill) for Gastrointestinal Transit Time Measures in Patients With Functional Gastrointestinal Symptoms and Dysmotility
Brief Title: Comparison of the Atmo Motility Gas Capsule System to the Reference Standard
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Atmo Biosciences Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A0015
Record Dates: First submitted 2023-01-24; First posted 2023-02-08 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Gastroparesis; Slow Transit Constipation; IBS
MeSH Terms: conditions — Gastroparesis | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: All participants will ingest the investigational and predicate device in a tandem ingestion. The order of device ingestion will be randomized, controlled centrally via an Electronic Data Capture system.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- SmartPill Monitoring System (Active Comparator): The SmartPill GI Monitoring System (Medtronic) offers a method for measuring gastric emptying time (GET), small bowel transit time (SBTT), colonic transit time (CTT), small bowel large bowel transit time (SLBTT) and whole gut transit time (WGTT) with a single test, which can be used as an aid for the diagnosis of both gastroparesis and slow transit constipation.
  The SmartPill System measures pH, temperature and pressure. It is approved for use in the measurement of GI transit times by the FDA.
  Interventions: Device: SmartPill Monitoring System
- Atmo Motility Gas Capsule System (Experimental): The Atmo Motility Gas Capsule System (Atmo Biosciences) offers a novel method for measuring GET, SBTT, SLBTT, CTT and WGTT. This device measures temperature, relative humidity, hydrogen concentration and carbon dioxide concentration, along with indicators of fermentation activity, capsule tumble and antenna reflectance as it transit through the GI tract.
  It has the added benefit of recording information on the fermentation and gas profiles within the GI tract.
  Interventions: Device: Atmo Motility Gas Capsule System

INTERVENTIONS:
Device: Atmo Motility Gas Capsule System — The Atmo System measures whole gut and regional gut transit times. Measurements of GI tract transit times are used for evaluating motility disorders.
  Gastric emptying time (GET) is indicated for the evaluation of patients with suspected gastroparesis. Delayed GET is implicated in such disorders as idiopathic and diabetic gastroparesis and functional non-ulcer dyspepsia.
  Colonic transit time (CTT) is indicated for the evaluation of colonic transit in patients with chronic constipation, to aid in differentiating slow and normal transit constipation. In the case where ileocecal junction transit cannot be determined the system will report combined Small and Large Bowel Transit Time (SLBTT).
  Transit times are derived from measures of temperature, relative humidity, hydrogen concentration, and carbon dioxide concentration, in conjunction with indicators of fermentation activity, capsule tumble, and antenna reflectance. Not for use in pediatric patients.
  Arms: Atmo Motility Gas Capsule System
Device: SmartPill Monitoring System — The SmartPill GI Monitoring System (Medtronic) offers a method for measuring gastric emptying time (GET), small bowel transit time (SBTT), colonic transit time (CTT), small bowel large bowel transit time (SLBTT) and whole gut transit time (WGTT) with a single test, which can be used as an aid for the diagnosis of both gastroparesis and slow transit constipation.
  The SmartPill System measures pH, temperature and pressure. It is approved for use in the measurement of GI transit times by the FDA.
  Arms: SmartPill Monitoring System

SUMMARY:
The study objective is to demonstrate the equivalence of the Atmo Motility Gas Capsule System with the predicate SmartPill in measuring gastric emptying time and colonic transit time through examination of device agreement.

DETAILED DESCRIPTION:
The clinical protocol for the study is designed to compare the performance of the Atmo Motility Gas Capsule System to the predicate device, the SmartPill GI Monitoring System, in patients with chronic GI symptoms suggestive of GI motility disorders (specifically gastroparesis and slow transit constipation), in order to demonstrate substantial equivalence. This study will involve the recruitment of symptomatic participants from a population that is representative of that for which the device is intended.

The primary objective of this study is the assessment of the agreement of Atmo Motility and SmartPill Systems' results with regards to both GET and CTT. The SmartPill is the accepted gold standard test for GI motility transit time analysis. Device agreement will be primarily examined through Bland-Altman analyses for GET and CTT measurements from the Atmo Motility and SmartPill Systems.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (M/F/other) between the ages of 22-80 years of age
2. High probability of compliance and completion of study.
3. Fulfilling one or more of the following criteria:

   A. Received a delayed gastric emptying result from a gastric emptying study (gastric scintigraphy [GES] or gastric emptying breath test [GEBT] or SmartPill) in the last two years AND/OR presenting with 2 or more of the following symptoms or signs: i. Nausea, vomiting, or retching (dry heaves) ii. Postprandial fullness or early satiety iii. Bloating or visible abdominal distention iv. Postprandial discomfort or pain AND/OR; B. Suffering from symptoms of chronic idiopathic constipation based on ROME IV criteria (exclusion of constipation caused by structural abnormalities), participant should have at least 1 bowel motion per week (either assisted or unassisted by medication) AND/OR; C. Suffering from symptoms of IBS-C based on ROME IV criteria
4. Participant or their legally authorized representative has the ability to provide informed consent and comply with the protocol.

Exclusion Criteria:

1. Recent abdominal and/or pelvic surgery (past 3 months)
2. Acute diverticulitis, confirmed by CT scan in past 3 months, diverticular stricture, and other intestinal strictures
3. Chronic daily use of nonsteroidal anti-inflammatory drugs (e.g. ibuprofen, naproxen)
4. Pregnant or breastfeeding
5. Patients on long-acting glucagon-like peptide (GLP-1)
6. Active implantable devices (e.g. gastric stimulator, pacemaker, defibrillator) [continuous glucose monitors are permitted]
7. Evidence of metabolic disease within the last six months (overt hypothyroidism [high TSH, low FT4], uncontrolled diabetes [hemoglobin A1c >10%] within the past 6 months) not stabilized within the past 3 months via constant medication (dosage and type must be consistent) usage
8. History of gastric bezoar formation
9. Presence of fistulas or other mechanical GI obstruction
10. Radiation enteritis
11. History of fecal impaction
12. Suspicion of other organic GI disease
13. Suspicion of obscure GI bleeding
14. Unable to stop medications that may alter gastric pH (such as proton pump inhibitors) for 7 days prior to and during study
15. Unable to stop medications that may alter GI motility (GLP-1 agonists, anticholinergics, metformin, antispasmodic, prokinetics) for 72 hours prior to and during study.
16. Chronic daily use of cannabinoids (e.g., dronabinol, marijuana)
17. Unable to stop laxatives (docusate, lactulose, sorbitol, senna, bisacodyl), suppositories (glycerin), and enema 72 hours prior to and during the study. Limited use of rescue laxatives is permissible at the investigators discretion but must be tracked in the electronic case report form (eCRF).
18. May require an MRI scan during the duration of this study
19. BMI > 40kg/m2
20. Allergies to any of the ingredients used in the standardized meal

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
GET as measured by the Atmo Motility System | Day 1 to Day 10
  Interpretation of gastric emptying time by central readers using the Atmo Motility System
GET as measured by the SmartPill System | Day 1 to Day 10
  Interpretation of gastric emptying time by central readers of the SmartPill System
CTT as measured by the Atmo Motility System | Day 1 to Day 10
  Interpretation of colonic transit time by central readers using the Atmo Motility System
CTT as measured by the SmartPill System | Day 1 to Day 10
  Interpretation of colonic transit time by central readers using the SmartPill System

SECONDARY OUTCOMES:
Classification as delayed or not for GI transit times: SBTT, OCTT, SLBTT and WGTT as determined by Atmo Motility System | Day 1 to Day 10
  Classification of all gut transit times as either delayed or not as measured by the Atmo System
Classification as delayed or not for GI transit times: SBTT, OCTT, SLBTT and WGTT as determined by SmartPill | Day 1 to Day 10
  Classification of all gut transit times as either delayed or not as measured by SmartPill
Classification as rapid or not for all transit times: GET, SBTT, OCTT, SLBTT, CTT and WGTT as determined by the Atmo Motility System | Day 1 to Day 10
  Classification of all gut transit times as either rapid or not as measured by Atmo
Classification as rapid or not for all transit times: GET, SBTT, OCTT, SLBTT, CTT and WGTT as determined by SmartPill | Day 1 to Day 10
  Classification of all gut transit times as either rapid or not as measured by SmartPill
Continuous transit time measures for SBTT, OCTT, SLBTT and WGTT for SmartPill and Atmo Motility Systems | Day 1 to Day 10
  Measurement of gut transit times as as measured by the SmartPill and Atmo Systems, expressed in hours:minutes
Qualitative description of per participant hydrogen and carbon dioxide gas profiles as determined by the Atmo Motility System | Day 1 to Day 10
  Description of gas production profiles as measured by the Atmo Motility System
Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), Serious Adverse Device Effects (SADEs), Unanticipated Serious Adverse Device Effects (USADEs) and device deficiencies | Day 0 to Day 31
  Description, number and outcomes of all adverse events, serious adverse events and others, summarized by recruitment site

CONTACTS AND LOCATIONS:
Overall Officials: Braden Kuo, MD, Principal Investigator — Massachusetts General Hospital; William Chey, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo B, Lee AA, Abell T, Attaluri A, Cline M, Hasler W, Ho V, Lembo AJ, Masoud A, McCallum R, Moshiree B, Quigley EMM, Rao SSC, Stocker A, Sanchez M, Sarosiek I, Surjanhata B, Zhou J, Chey WD. The Assessment of Gastrointestinal Transit by the Atmo Capsule: A Comparison With the SmartPill Capsule. Clin Gastroenterol Hepatol. 2025 Aug;23(9):1633-1641.e8. doi: 10.1016/j.cgh.2024.12.013. Epub 2025 Jan 30. PMID 39889900